CLINICAL TRIAL: NCT01393782
Title: Intravenous AII for the Treatment of Severe Hypotension in High Output Shock: A Pilot Study
Acronym: ATHOS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 111016
Record Dates: First submitted 2011-07-12; First posted 2011-07-13 (Estimated); Results first posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2023-10

CONDITIONS: Septic Shock
Keywords: high output shock; distributive shock; warm shock; septic shock; pressor; angiotensin; ATII; vasopressor
MeSH Terms: conditions — Shock, Septic | interventions — Angiotensin II

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Angiotensin (Active Comparator): The angiotensin arm will receive angiotensin II acetate at an initial dose of 20ng/kg/min, titratable during the study (6 hours) for mean arterial pressure (MAP) goals as outlined in the protocol.
  Interventions: Drug: Angiotensin II
- Control (Placebo Comparator): Control patients will receive placebo intravenously equal in duration, color and volume to the intervention arm's angiotensin II.
  Interventions: Drug: Angiotensin II

INTERVENTIONS:
Drug: Angiotensin II — All patients will have their vasopressors titrated to a mean arterial pressure (MAP) of 65 mm of Hg (standard MAP goal in the ICU for patients suffering from shock). Patients will then be randomized to control or IV AII. In the interventional arm, AII will start at a dose of 20ng/kg/min; the dose can then be titrated up to 30ng/kg/min, and then to 40ng/kg/min. The intervention will last for 6 hours. Each patient will start with the assigned starting dose indicated above. After the first hour, if the patient is still requiring standing norepinephrine (the standard vasopressor for the treatment of shock in the GW ICU), the dose of the control/interventional drug can be increased 50%. After the second hour, if the patient is still requiring a standing dose of norepinephrine, the control/interventional can be increased again to twice the initial dose. At the end of 6 hours, the study drug will be titrated off.

SUMMARY:
The investigators propose a dose finding study to determine the feasibility of Angiotensin II (AII) to increase mean arterial pressure in high-output shock. If AII can be shown to increase mean arterial pressure, this could lead to future pharmacologic development based on the AII hormonal pathway. The investigators propose a 20 patient, randomized, placebo-controlled, blinded study in the treatment of high-output shock. Patients with high-output shock and a cardiovascular SOFA (sequential organ failure score) score of > 4 will be eligible. In addition, patients must already be receiving cardiac output monitoring and have a cardiac index > 2.4 L/min/ 1.73 m2. Patients will be randomized to intravenous AII or saline in a blinded fashion. There will be 10 patients in each arm. This is a safety and dose finding feasibility study. The investigators are starting with a small cohort consistent with similar types of studies. The investigators estimate that ten patients in each arm will generate a basis for determining if there is sufficient signal for AII to improve blood pressure at the doses outlined. The primary endpoint in the study will be the effect of AII on the standing dose of norepinephrine which is required to maintain a mean arterial pressure (MAP) of 65 mmHg. Secondary endpoints will be the effect of AII on urine output, serum lactate, and creatinine clearance. 30 day post dose mortality will also be assessed. Subjects discharged prior to day 30 will be contacted by telephone for this assessment.

ELIGIBILITY:
Inclusion Criteria:

1. High-output shock
2. Cardiovascular SOFA score of > 4
3. Cardiac Index > 2.4 liters/min/BSA 1.73m2
4. Indwelling arterial line already present as part of standard care
5. Age > 21 years of age
6. Signed consent form
7. Use of indwelling urinary catheter as standard care expected at least for 12 hours during the study interventions

Exclusion Criteria:

1. Patients with acute coronary syndrome
2. Patients with a known history of vasospasm
3. Patients with a history of asthma
4. Patients currently experiencing bronchospasm
5. Patients with active bleeding with an anticipated need for > 4 units of PRBC or Hemoglobin < 7g/dL or any other condition that would contraindicate drawing serial blood samples

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lakhmir Chawla, MD, Principal Investigator — GW University
Locations (1):
- GW University, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Chawla LS, Busse L, Brasha-Mitchell E, Davison D, Honiq J, Alotaibi Z, Seneff MG. Intravenous angiotensin II for the treatment of high-output shock (ATHOS trial): a pilot study. Crit Care. 2014 Oct 6;18(5):534. doi: 10.1186/s13054-014-0534-9. PMID 25286986

RESULTS

PARTICIPANT FLOW:
Groups:
- Angiotensin: The angiotensin arm will receive angiotensin II acetate at an initial dose of 20ng/kg/min, titratable during the study (6 hours) for MAP goals as outlined in the protocol.
Period: Overall Study
Arm/Group | Angiotensin | Control
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Angiotensin | Control | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (17.5) | 57.3 (12.4) | 62.9 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 6 | 9 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 6 | 3 | 9
  Black | 3 | 5 | 8
  Other | 1 | 2 | 3
Baseline Sequential Organ Failure Assessment (SOFA) score, Continous [Mean (Standard Deviation); unit: Scores on a scale 0-24 (higher is worse)] | 14.9 (2.8) | 16.9 (2.9) | 15.9 (3.0)
Acute physiology and chronic health evaluation (APACHE) score, continous [Mean (Standard Deviation); unit: Scores on a scale 0-71 (higher is worse)] | 27.2 (9.7) | 34 (6.8) | 30.6 (8.9)
Ischemic heart disease [Count of Participants; unit: Participants] | 1 | 1 | 2
Congestive heart failure [Count of Participants; unit: Participants] | 2 | 0 | 2
Chronic obstructive pulmonary disease [Count of Participants; unit: Participants] | 2 | 0 | 2
Diabetes [Count of Participants; unit: Participants] | 4 | 3 | 7
Chronic kidney disease [Count of Participants; unit: Participants] | 3 | 4 | 7
Hemodialysis [Count of Participants; unit: Participants] | 0 | 1 | 1
Liver disease [Count of Participants; unit: Participants] | 5 | 4 | 9
Cancer [Count of Participants; unit: Participants] | 1 | 5 | 6
Immunocompromised state (as defined by steroid therapy or history of immunocompromise disease) [Count of Participants; unit: Participants] | 1 | 5 | 6
Steroids [Count of Participants; unit: Participants] | 1 | 2 | 3
Hypertension [Count of Participants; unit: Participants] | 4 | 5 | 9
Cerebrovascular accident [Count of Participants; unit: Participants] | 4 | 1 | 5
Acute kidney injury [Count of Participants; unit: Participants] | 9 | 8 | 17
Baseline Norepinephrine dose [Mean (Standard Deviation); unit: mcg/min] | 19.8 (11.7) | 30.3 (20.4) | 25.1 (17.0)
Baseline Vasopressin dose [Mean (Standard Deviation); unit: units/min] | 0.03 (0.02) | 0.05 (0.02) | 0.04 (0.02)

OUTCOME MEASURES:

1. Primary Outcome: Standing Dose of Norepinephrine Which is Required to Maintain a Mean Arterial Pressure (MAP) of 65 mmHg - Hour 1
Description: The primary endpoint in the study will be the effect of AII on the standing dose of norepinephrine which is required to maintain a mean arterial pressure (MAP) of 65 mmHg.
Time Frame: 1 hour after initiation of angiotensin II (ATII)
Measure: Mean (Standard Deviation); unit: mcg/min
Arm/Group | Angiotensin | Control
Number analyzed (Participants) | 10 | 10
mcg/min | 7.4 (12.4) | 27.6 (29.3)

2. Primary Outcome: Standing Dose of Norepinephrine Which is Required to Maintain a MAP of 65 mmHg - Hour 2
Description: The primary endpoint in the study will be the effect of AII on the standing dose of norepinephrine which is required to maintain a MAP of 65 mmHg.
Time Frame: 2 hours after initiation of ATII
Measure: Mean (Standard Deviation); unit: mcg/min
Arm/Group | Angiotensin | Control
Number analyzed (Participants) | 10 | 10
mcg/min | 7.3 (11.9) | 28.6 (30.2)

3. Secondary Outcome: Mortality
Description: 30 day post dose mortality will be assessed. Subjects discharged prior to day 30 will be contacted by telephone for this assessment.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Angiotensin | Control
Number analyzed (Participants) | 10 | 10
Participants | 5 | 6

ADVERSE EVENTS:
Arm/Group | Angiotensin | Control
All-Cause Mortality (participants affected / at risk) | 5/10 | 6/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 2/10 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Angiotensin (N=10) | Control (N=10)
Hypertension (Cardiac disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes